CLINICAL TRIAL: NCT00480519
Title: Use of Sedation and Local Anesthesia in Meatotomy: A Prospective Comparison Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Schneider Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: scmc4304ctil
Record Dates: First submitted 2007-05-30; First posted 2007-05-31 (Estimated); Last update posted 2007-05-31 (Estimated); Status verified 2007-05

CONDITIONS: Pain
Keywords: meatotomy; meatal stenosis; local anaesthesia; feasibility; pain control
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Meatotomy

SUMMARY:
The aim of the study is to prospectively investigate the feasibility, pain control, and outcome of meatotomy performed under sedation and local anaesthesia compared with general anaesthesia with and without patient block

DETAILED DESCRIPTION:
Background- Meatal stenosis requiring surgery occurs more often in circumcised than in uncircumcised boys, with an estimated rate of 7.3%. At our institute, meatotomy is usually performed under general anesthesia and penile block is routinely added after induction. Recently, several reports have described the performance of meatotomy as an office procedure under local anesthesia, with good patient tolerability and a considerable reduction in operative time and costs.

Purpose - The aim of the study is to prospectively investigate the feasibility, pain control, and outcome of meatotomy performed under sedation and local anaesthesia compared with general anaesthesia with and without patient block.

Materials and Methods- The study population will include 75 otherwise healthy boys aged 3 years to 15 years scheduled for meatotomy at our institute. Children with ASA grade >2 will be excluded. The children will be reexamined by a senior pediatric ulologist to confirm the need for surgery. All children and their parents will be given a detailed explanation of the procedure and of the anesthesia and pain control options available by a urology nurse, pediatric urologist, and anesthesist.

Prior to surgery, study participants will be randomly allocated to one of the following groups:

Group 1 will include 25 patients who will undergo meatotomy under sedation and local anesthesia. The penis will be topically treated with EMLA cream one hour before surgery and then covered with tegaderm. In children aged 3-5 years, sedation will consist of midazolam 0.5 mg/kg (up to 10 mgs) p.o., administered 20 minutes before surgery; children aged 5 years and older will receive nitrous oxide (up to 60%) with oxygen. All patients will be connected to a pulse oximeter and monitored by a sedation nurse or an anesthesist.

Group 2 will include 25 boys operated on under general anaesthesia. Anesthesia will be induced by Sevoflurane 8% or IV propofol 2 mg/kg and maintained with sevoflurane 3% or isoflurane 1% and nitrous oxide. Ropivacaine 0.2% 1 cc-5 cc will be administered for penile block following induction.

Group 3 will include 25 boys operated on under general anesthesia, like group 2, but without penile block.

All children in all groups will receive paracetamol 15 mg/kg (up 500 mg) as suppository or suspension after completion of the meatotomy, and will be monitored by a sedation nurse until they are fully recovered. They will be discharged from the hospital after a successful spontaneous void.

Prior to patient discharge, the parents will be asked to complete a form grading their child's current pain level and their general satisfaction with the procedure (Appendix I). Boys older than 5 years will be asked to complete their own pain scale as well.

Twenty-four hours after surgery, the parents will be asked, by telephone, to again grade their child's current pain; to report the type and doses of pain medications used within this time frame, to score their child's voiding quality; and to rate their general satisfaction (Appendix II).

All patients will be invited for a follow-up visit at the clinic one month after the procedure. At that time, a urologist will assess the meatal width and voiding quality (Appendix III).

ELIGIBILITY:
Inclusion Criteria:

* Boys between 3 years and 18 years with meatal stenosis requiring meatotomy

Exclusion Criteria:

* ASA grade > 2

Ages: 3 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2007-05; Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
pain control, voiding quality | one month after the procedure

SECONDARY OUTCOMES:
general satisfaction | before the child is discharged from the hospital, and one month after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: David Ben-Meir, MD, Principal Investigator — Schneider Chlidren's medical Center of Israel
Locations (1):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel